CLINICAL TRIAL: NCT03887013
Title: Cardiac Metabolic Modulator Treatment for Improvement of Left Ventricular Diastolic Function in Patients With Coronary Heart Disease: a Prospective, Randomized Controlled Study
Brief Title: Cardiac Metabolic Modulator Treatment for Improvement of Diastolic Function in Patients With Coronary Heart Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFH20180050
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2018-10

CONDITIONS: Coronary Heart Disease; Diastolic Dysfunction
MeSH Terms: conditions — Coronary Disease | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHD routine therapy (No Intervention): Patients with CHD will be treated with evidence-based therapy including antiplatelet drugs,beta-blockers,statins,angiotensin-converting enzyme inhibitor (ACEI),nitrates,etc. Percutaneous coronary intervention (PCI) could be performed if needed.
- CHD routine therapy+Trimetazidine (Experimental): Apart from the drug and PCI therapy mentioned above,patients will be given treatment of trimetazidine.
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — Trimetazidine is given as 20mg every time and three times per day (Tid) or 20mg every time and two times per day (when renal function is declined).
  Other Names: Cardiac metabolic modulator
  Arms: CHD routine therapy+Trimetazidine

SUMMARY:
Based on accumulating evidence showing that impaired cardiac energetic metabolism plays important role in the mechanism of cardiac diastolic dysfunction,the study is designed to evaluate whether metabolic modulator treatment with trimetazidine could have beneficial effects on patients with coronary heart disease(CHD) and ventricular diastolic dysfunction.This study is a prospective,randomised,open-label trial to assess the efficacy of trimetazidine treatment in improving diastolic function in CHD patients with diastolic dysfunction.

DETAILED DESCRIPTION:
The primary objective of this trial is to determine whether the 24-week trimetazidine therapy, as an adjunct to routine treatment for CHD, would improve diastolic function in patients with ischemic heart disease compared to the routine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50 and 79 years,male or female (without pregnancy).
* Diagnosed CHD by coronary angiography,with stenoses in main bifurcations less than 70% after PCI treatment.
* Left ventricular ejection fraction(LVEF) more than 50% assessed by ultracardiography.
* Characteristics of diastolic dysfunction by ultracardiography (more than 2 criteria as following):(1)Average E/e'>14,(2)Septal e' velocity <7 cm/s or lateral e' velocity <10 cm/s,(3)Tricuspid regurgitation (TR) velocity >2.8m/s,(4)Left atrium (LA) volume index >34ml/m2.
* Not yet being treated by trimetazidine.
* Provided informed consent.

Exclusion Criteria:

* Acute heart failure or acute exacerbation of chronic heart failure.
* LVEF less than 50% at admission or in the past.
* History of malignant tumor or life expectancy under 12 months.
* Acute myocardial infarction or unstable angina pectoris within 3 months.
* Scheduled coronary artery bypass grafting therapy within 6 months.
* Diagnosed or considered valvular heart disease, hypertrophic cardiomyopathy,restrictive cardiomyopathy or pericardium diseases.
* Significant hepatic impairment (Serum glutamate-pyruvate transaminase more than 3 times normal upper limit) or severe renal dysfunction (eGFR≤30 ml/min/1.73m2).
* Known or considered Parkinson's Disease.
* Known hypersensitivity or intolerance to trimetazidine.
* Pregnancy and lactation period.
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol.
* Participation in another clinical trial within the past 30 days.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2019-03-25 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Percentage difference of patients with II or III degree diastolic dysfunction in each arm | Within 6 months after patients being enrolled
  II or III degree diastolic dysfunction is defined as average E/e' ratio more than 10

SECONDARY OUTCOMES:
Average E/e' ratio change between week 24 and baseline | Within 6 months after patients being enrolled
  Average e/e' is evaluated by ultracardiography
E' velocity change of septum or of left ventricular lateral wall in m/s between week24 and baseline | Within 6 months after patients being enrolled
  E' velocity change of septum or of left ventricular lateral wall is evaluated by ultracardiography
Velocity of tricuspid regurgitation change in m/s between week 24 and baseline | Within 6 months after patients being enrolled
  Velocity of tricuspid regurgitation is evaluated by ultracardiography
Index of left atrium volume change between week 24 and baseline | Within 6 months after patients being enrolled
  Index of left atrium volume is evaluated by ultracardiography
Concentration of the plasma N-terminal pro-B-type natriuretic peptide (NT-proBNP) change in pg/ml between week 24 and baseline | Within 6 months after patients being enrolled
  NT-proBNP is tested by Fuwai Hospital laboratory
Number of participants with cardiovascular death and being rehospitalized for heart failure within 24 weeks treatment | Within 6 months after patients being enrolled
  This number will be acquired during follow up
Concentration of glycated hemoglobin (HbA1c) change in patients with diabetes mellitus (DM) between week 24 and baseline | Within 6 months after patients being enrolled
  HbA1c (%)is tested by Fuwai Hospital laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhao, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China